CLINICAL TRIAL: NCT07226245
Title: Evaluating Pharmacokinetics of Three Methadone Dosing Strategies During Cardiac Surgery With Cardiopulmonary Bypass
Brief Title: Methadone Pharmacokinetics in Cardiac Surgery
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00136746
Record Dates: First submitted 2025-11-04; First posted 2025-11-10 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-09

CONDITIONS: Postoperative Pain Management
Keywords: methadone pharmacokinetics; cardiac surgery; pain management; cardiac surgery recovery; methadone
MeSH Terms: conditions — Agnosia | interventions — Methadone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Single dose of methadone (Active Comparator): Single dose of methadone administered at induction of anesthesia
  Interventions: Drug: Single dose of methadone
- Split dose of methadone (Experimental): Split dose of methadone post cardiopulmonary bypass
  Interventions: Drug: Split dose of methadone
- Balanced split dose of methadone (Experimental): Balanced split dose of methadone post cardiopulmonary bypass
  Interventions: Drug: Balanced split dose of methadone

INTERVENTIONS:
Drug: Single dose of methadone — Single dose of methadone 0.3 mg/kg actual body weight (max 30 mg) administered at induction of anesthesia
  Arms: Single dose of methadone
Drug: Split dose of methadone — Split dose of methadone 0.2 mg/kg actual body weight at induction and 0.1 mg/kg actual body weight post cardiopulmonary bypass
  Arms: Split dose of methadone
Drug: Balanced split dose of methadone — Balanced split dose of methadone 0.15 mg/kg actual body weight at induction and 0.15 mg/kg actual body weight post cardiopulmonary bypass
  Arms: Balanced split dose of methadone

SUMMARY:
Cardiac surgery frequently leads to significant postoperative pain, with multiple different drug regimens being utilized (both opioid and non-opioid) in an attempt to alleviate this surgical pain. Methadone is currently one of the drugs that is being utilized to help control the pain. It can be given during and/or after surgery. This study hopes to identify the optimal dose of methadone to use to treat this surgical pain.

DETAILED DESCRIPTION:
The uncertainty regarding optimal methadone dosing and the necessity of post-cardiopulmonary bypass (CPB) supplementation provides a compelling rationale for this study. Specifically, it remains unknown whether a single higher initial dose of methadone can adequately maintain analgesic plasma concentrations throughout cardiac surgery and recovery, or if a split-dosing strategy administering a lower initial dose followed by an additional dose post-CPB might offer similar or improved analgesic outcomes with fewer side effects. This study will evaluate pharmacokinetics of methadone using three different dosing strategies in patients undergoing cardiac surgery with CPB.

ELIGIBILITY:
Inclusion Criteria:

* Elective cardiac surgery requiring median sternotomy and cardiopulmonary bypass (CABG, valve, combined CABG/valve surgeries)
* Anticipated extubation within 12 hours postoperatively
* No prior opioid use within 30 days of surgery
* Ability to provide informed consent

Exclusion Criteria:

* Severe liver or kidney dysfunction (Child-Pugh class B/C, eGFR <30 mL/min/1.73m², creatinine >2 mg/dL, dialysis)
* Allergy to methadone or fentanyl
* Use of CYP3A4 inducers (rifampin, phenytoin, carbamazepine), CYP3A4 inhibitors (ketoconazole, erythromycin, clarithromycin, itraconazole), SSRIs (fluoxetine, sertraline, paroxetine, citalopram, escitalopram, fluvoxamine)
* Body mass index >40 kg/m²
* Corrected QT interval interval >500 milliseconds
* Intubation anticipated >12 hours
* History of illicit drug use or alcohol or opioid abuse use disorder within last 12 months
* Mechanical circulatory support, heart transplant, deep hypothermic circulatory arrest procedures
* Left Ventricular Ejection Fraction <30%
* Pulmonary disease requiring oxygen therapy
* Preoperative inotropic support or intra-aortic balloon pump
* Emergency surgery
* Postoperative regional anesthesia
* Hemofiltration during cardiopulmonary bypass

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Plasma methadone concentration (ng/mL) 10 min post initial dose | 10 minutes
  Plasma methadone concentration will be measured 10 minutes post initial methadone dose
Plasma methadone concentration (ng/mL) 30 min post initial dose | 30 minutes
  Plasma methadone concentration will be measured 30 minutes post initial methadone dose pre cardiopulmonary bypass
Plasma methadone concentration (ng/mL) 60 min post initial dose | 60 minutes
  Plasma methadone concentration will be measured 60 minutes post initial methadone dose pre cardiopulmonary bypass
Plasma methadone concentration (ng/mL) 10 min post start of cardiopulmonary bypass | 10 minutes
  Plasma methadone concentration will be measured 10 minutes after cardiopulmonary bypass started
Plasma methadone concentration (ng/mL) 30 min post start of cardiopulmonary bypass | 30 minutes
  Plasma methadone concentration will be measured 30 minutes after cardiopulmonary bypass started
Plasma methadone concentration (ng/mL) 60 min post start of cardiopulmonary bypass | 60 minutes
  Plasma methadone concentration will be measured 60 minutes after cardiopulmonary bypass started
Plasma methadone concentration (ng/mL) 10 min post cardiopulmonary bypass completion | 10 minutes
  Plasma methadone concentration will be measured 10 minutes after cardiopulmonary bypass ended
Plasma methadone concentration (ng/mL) 120 min post start of cardiopulmonary bypass | 120 minutes
  Plasma methadone concentration will be measured 120 minutes after cardiopulmonary bypass started
Plasma methadone concentration (ng/mL) before first analgesic request | up to 72 hours
  Plasma methadone concentration will be measured at the time of first analgesic request by participant
Plasma methadone concentration (ng/mL) 3 hours post Intensive Care Unit arrival | 3 hours
  Plasma methadone concentration will be measured 3 hours post Intensive Care Unit arrival
Plasma methadone concentration (ng/mL) 12 hours post Intensive Care Unit arrival | 12 hours
  Plasma methadone concentration will be measured 12 hours post Intensive Care Unit arrival
Plasma methadone concentration (ng/mL) 24 hours post Intensive Care Unit arrival | 24 hours
  Plasma methadone concentration will be measured 24 hours post Intensive Care Unit arrival

SECONDARY OUTCOMES:
pain intensity score | 2, 4, 8, 12, 24, 48, and 72 hours postoperatively and month 3
  Pain intensity score will be measured using the visual analog scale. Scores will be measured on a scale of 0-10, with 0=no pain and 10=most severe pain
patient global impression of change | 24, 48, and 72 hours after removal of the breathing tube
  Patient Global Impression of Change will be used to assess patient-perceived analgesic effectiveness and overall postoperative recovery. Total score range is 1-7 with a higher score indicating considerable improvement with treatment.
postoperative opioid consumption | up 72 hours postop
  total postoperative opioid consumption in morphine milligram equivalents
duration of postoperative mechanical ventilation | up to 72 hours postop
  number of minutes with postoperative mechanical ventilation
time of ambulation | up to 48 hours postop
  number of minutes until patient first ambulates after surgery
length of Intensive Care Unit stay | up to 3 days postop
  number of hours spent in Intensive Care Unit
length of hospital length stay | up to 7 days postop
  number of days spent in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Ettore Crimi, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
study results will be shared instead of individual patient data